CLINICAL TRIAL: NCT05252676
Title: Evaluation of Correlations Between Radiologic Features and Pathologic Subtypes of Ground Glass Opacity Featured Lung Adenocarcinoma Via Whole-Mount Section
Brief Title: Evaluation of Correlations Between Radiologic Features and Pathologic Subtypes of GGO LUAD Via WMS (ECTOP-1011)
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Professor, Fudan University
Other Study IDs: IRB2106237-23
Record Dates: First submitted 2022-02-13; First posted 2022-02-23 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Adenocarcinoma of Lung
Keywords: Ground glass opacity
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with ground glass opacity featured lung adenocarcinoma who are candidates for surgery.

SUMMARY:
This study is one of the Eastern Cooperative Thoracic Oncology Projects (ECTOP-1011). It aims to evaluate the correlations between radiologic features and pathologic subtypes of ground glass opacity featured lung adenocarcinoma via whole-mount section.

DETAILED DESCRIPTION:
The pathological lepidic growth pattern was believed to relate to the ground-glass component, whereas invasive adenocarcinoma patterns relate to the solid component. However, the solid components might be fibrosis rather tumor; and previous studies demonstrated the ground-glass components might be invasive lesions. Therefore, it is of considerable significance to establish the correlations between radiologic features and pathologic subtypes of ground glass opacity featured lung adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Ground glass opacity featured lung nodule diagnosed by thin-section computed tomography(TSCT)
* Pre-operation clinical IA stage
* Pulmonary lobectomy or segmentectomy
* Provision of informed consent

Exclusion Criteria:

* Postoperative diagnosis of non-adenocarcinoma or mucinous adenocarcinoma
* The surgical specimens fail to satisfy requirement of inflation and formalin fixation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: East Asian population
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of correlations between radiologic features and pathologic subtypes | about 14 days
  Evaluation of correlations between radiologic features and pathologic subtypes of ground glass opacity featured lung adenocarcinoma

SECONDARY OUTCOMES:
Specificity, Sensitivity, and Repeatability | about 14 days
  The specificity, sensitivity, and repeatability of invasiveness diagnosis based on the Whole-Mount Section

CONTACTS AND LOCATIONS:
Overall Officials: Haiquan Chen, M.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Noguchi M, Morikawa A, Kawasaki M, Matsuno Y, Yamada T, Hirohashi S, Kondo H, Shimosato Y. Small adenocarcinoma of the lung. Histologic characteristics and prognosis. Cancer. 1995 Jun 15;75(12):2844-52. doi: 10.1002/1097-0142(19950615)75:123.0.co;2-#. PMID 7773933
- [Background] Koike T, Terashima M, Takizawa T, Watanabe T, Kurita Y, Yokoyama A. Clinical analysis of small-sized peripheral lung cancer. J Thorac Cardiovasc Surg. 1998 May;115(5):1015-20. doi: 10.1016/S0022-5223(98)70399-X. PMID 9605069
- [Background] Suzuki K, Asamura H, Kusumoto M, Kondo H, Tsuchiya R. "Early" peripheral lung cancer: prognostic significance of ground glass opacity on thin-section computed tomographic scan. Ann Thorac Surg. 2002 Nov;74(5):1635-9. doi: 10.1016/s0003-4975(02)03895-x. PMID 12440622
- [Background] Suzuki K, Kusumoto M, Watanabe S, Tsuchiya R, Asamura H. Radiologic classification of small adenocarcinoma of the lung: radiologic-pathologic correlation and its prognostic impact. Ann Thorac Surg. 2006 Feb;81(2):413-9. doi: 10.1016/j.athoracsur.2005.07.058. PMID 16427823
- [Background] Travis WD, Asamura H, Bankier AA, Beasley MB, Detterbeck F, Flieder DB, Goo JM, MacMahon H, Naidich D, Nicholson AG, Powell CA, Prokop M, Rami-Porta R, Rusch V, van Schil P, Yatabe Y; International Association for the Study of Lung Cancer Staging and Prognostic Factors Committee and Advisory Board Members. The IASLC Lung Cancer Staging Project: Proposals for Coding T Categories for Subsolid Nodules and Assessment of Tumor Size in Part-Solid Tumors in the Forthcoming Eighth Edition of the TNM Classification of Lung Cancer. J Thorac Oncol. 2016 Aug;11(8):1204-1223. doi: 10.1016/j.jtho.2016.03.025. Epub 2016 Apr 21. PMID 27107787
- [Background] Lim HJ, Ahn S, Lee KS, Han J, Shim YM, Woo S, Kim JH, Yie M, Lee HY, Yi CA. Persistent pure ground-glass opacity lung nodules >/= 10 mm in diameter at CT scan: histopathologic comparisons and prognostic implications. Chest. 2013 Oct;144(4):1291-1299. doi: 10.1378/chest.12-2987. PMID 23722583
- [Background] Suzuki K, Koike T, Asakawa T, Kusumoto M, Asamura H, Nagai K, Tada H, Mitsudomi T, Tsuboi M, Shibata T, Fukuda H, Kato H; Japan Lung Cancer Surgical Study Group (JCOG LCSSG). A prospective radiological study of thin-section computed tomography to predict pathological noninvasiveness in peripheral clinical IA lung cancer (Japan Clinical Oncology Group 0201). J Thorac Oncol. 2011 Apr;6(4):751-6. doi: 10.1097/JTO.0b013e31821038ab. PMID 21325976
- [Background] Son JY, Lee HY, Lee KS, Kim JH, Han J, Jeong JY, Kwon OJ, Shim YM. Quantitative CT analysis of pulmonary ground-glass opacity nodules for the distinction of invasive adenocarcinoma from pre-invasive or minimally invasive adenocarcinoma. PLoS One. 2014 Aug 7;9(8):e104066. doi: 10.1371/journal.pone.0104066. eCollection 2014. PMID 25102064
- [Background] Thunnissen E, Beasley MB, Borczuk AC, Brambilla E, Chirieac LR, Dacic S, Flieder D, Gazdar A, Geisinger K, Hasleton P, Ishikawa Y, Kerr KM, Lantejoul S, Matsuno Y, Minami Y, Moreira AL, Motoi N, Nicholson AG, Noguchi M, Nonaka D, Pelosi G, Petersen I, Rekhtman N, Roggli V, Travis WD, Tsao MS, Wistuba I, Xu H, Yatabe Y, Zakowski M, Witte B, Kuik DJ. Reproducibility of histopathological subtypes and invasion in pulmonary adenocarcinoma. An international interobserver study. Mod Pathol. 2012 Dec;25(12):1574-83. doi: 10.1038/modpathol.2012.106. Epub 2012 Jul 20. PMID 22814311
- [Background] Isaka T, Yokose T, Ito H, Imamura N, Watanabe M, Imai K, Nishii T, Woo T, Yamada K, Nakayama H, Masuda M. Comparison between CT tumor size and pathological tumor size in frozen section examinations of lung adenocarcinoma. Lung Cancer. 2014 Jul;85(1):40-6. doi: 10.1016/j.lungcan.2014.03.023. Epub 2014 Apr 1. PMID 24751107